CLINICAL TRIAL: NCT03125603
Title: Census and Follow-up of the Side Effects in the New Immunotherapeutic Treatments Anti-PD-(L)-1 and Anti-CTLA-4 of the Non Small Cells Lung Cancer
Brief Title: Side Effects of Anti-PD-(L)-1 and Anti CTLA-A4 in the Non Small Cells Lung Cancer
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Alexandre Niset, Med student, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: 2017/15MAR/137
Record Dates: First submitted 2017-04-13; First posted 2017-04-24 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Drug-Related Side Effects and Adverse Reactions
Keywords: Immunotherapy; Anti-PD-(L)-1; Anti-CTLA-4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC's patients: Patients with NSCLC treated in Cliniques Universitaires Saint-Luc with immunotherapy.
  Consultation of the patient's medical files at the hospital.
  Interventions: Other: Consultation of the patient's medical files at the hospital

INTERVENTIONS:
Other: Consultation of the patient's medical files at the hospital — Gradation of the adverse events according to CTCAE scale 4.03 (June 2010).

SUMMARY:
The immune-related adverse events (irAEs) linked to the important activation of the immune system by new immunotherapy treatments in patients affected by Non-small-cell lung carcinoma (NSCLC) have not received a lot of systematic study or been monitored over time outside of clinical trials.

This study aims to verify, on the basis of the data collected in a prospective and retrospective manner, that the side-effects due of anti-PD-(L)-1 or anti-CTLA-4 treatments observed in the target population of the controlled clinical trials are the same as in the general clinical population.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with NSCLC treated in Cliniques Universitaires Saint-Luc with immunotherapy in first or second line.

Exclusion Criteria:

* The refusal to sign the consent.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cliniques Universitaires Saint-Luc's patients with NSCLC eligible and treated with immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Census and monitor of the side-effects due to the immunotherapy treatment. | Through study completion, an average of 20 months.
  Census of the side-effect type, severity according to the CTCAE and monitoring the side-effect's development.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Pieters, MD, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Result] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Result] Michot JM, Bigenwald C, Champiat S, Collins M, Carbonnel F, Postel-Vinay S, Berdelou A, Varga A, Bahleda R, Hollebecque A, Massard C, Fuerea A, Ribrag V, Gazzah A, Armand JP, Amellal N, Angevin E, Noel N, Boutros C, Mateus C, Robert C, Soria JC, Marabelle A, Lambotte O. Immune-related adverse events with immune checkpoint blockade: a comprehensive review. Eur J Cancer. 2016 Feb;54:139-148. doi: 10.1016/j.ejca.2015.11.016. Epub 2016 Jan 5. PMID 26765102
- [Result] Villadolid J, Amin A. Immune checkpoint inhibitors in clinical practice: update on management of immune-related toxicities. Transl Lung Cancer Res. 2015 Oct;4(5):560-75. doi: 10.3978/j.issn.2218-6751.2015.06.06. PMID 26629425
- [Result] Postow MA, Callahan MK, Wolchok JD. Immune Checkpoint Blockade in Cancer Therapy. J Clin Oncol. 2015 Jun 10;33(17):1974-82. doi: 10.1200/JCO.2014.59.4358. Epub 2015 Jan 20. PMID 25605845
- [Result] Champiat S, Lambotte O, Barreau E, Belkhir R, Berdelou A, Carbonnel F, Cauquil C, Chanson P, Collins M, Durrbach A, Ederhy S, Feuillet S, Francois H, Lazarovici J, Le Pavec J, De Martin E, Mateus C, Michot JM, Samuel D, Soria JC, Robert C, Eggermont A, Marabelle A. Management of immune checkpoint blockade dysimmune toxicities: a collaborative position paper. Ann Oncol. 2016 Apr;27(4):559-74. doi: 10.1093/annonc/mdv623. Epub 2015 Dec 28. PMID 26715621
- [Result] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847